CLINICAL TRIAL: NCT00129480
Title: Improving the Treatment of Chronic Pain in Primary Care
Brief Title: Improving Chronic Pain Treatment in Primary Care
Acronym: SEACAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMI 03-195
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-01

CONDITIONS: Pain; Chronic Disease; Depression
Keywords: veterans; pain and chronic disease; disease management; depression; primary health care; practice guidelines; guideline adherence; narcotics; patient compliance; randomized controlled trial
MeSH Terms: conditions — Pain; Chronic Disease; Depression; Patient Compliance | interventions — Insemination, Artificial, Heterologous; Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Assistance with Pain Treatment (Experimental): Care management intervention including assessment, decision support, patient activation, education and followup, provider education, feedback to providers
  Interventions: Behavioral: Assistance with Pain treatment
- Treatment as usual (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Assistance with Pain treatment — Care management intervention including assessment, decision support, patient activation, education and followup, provider education, feedback to providers. Intervention delivered for 12 months.
  Arms: Assistance with Pain Treatment

SUMMARY:
The primary objective of this study is to determine to what extent a collaborative intervention improves chronic pain-related outcomes in a VA primary care setting. We will also determine to what extent the intervention affects 1) treatment of co-occurring depression, 2) adherence of providers to guidelines for treating chronic pain, and 3) patient and provider satisfaction and attitudes related to chronic pain treatment.

DETAILED DESCRIPTION:
Background:

Chronic pain is very common, and associated with substantial impairment and increased healthcare utilization. Implementation of treatment guidelines has been problematic, and chronic pain remains undertreated. Because of the prevalence of chronic pain among veterans, the VHA created a National Pain Management Strategy and adopted pain as the "5th vital sign."

Objectives:

Our primary objective was to determine to what extent a collaborative intervention improves chronic pain-related outcomes (pain-related function, pain severity and depression severity) in a VA primary care setting over six and 12 months. We also investigated to what extent the intervention affected 1) treatment of comorbid depression, 2) adherence of providers to guidelines for chronic pain, 3) patient and provider satisfaction and attitudes related to chronic pain treatment, and 4) incremental benefit (pain disability-free days) and incremental health services costs.

Methods:

The study was a cluster randomized controlled trial of a collaborative care intervention "Assistance with Pain Treatment" (APT) versus treatment as usual (TAU) at five primary care clinics of one Department of Veterans Affairs Medical Center.

401 patients and 42 primary care clinicians participated. APT included a 2-session clinician education program, patient assessment, education and activation, symptom monitoring, feedback and recommendations to clinicians and facilitation of specialty care. We randomized clinicians to APT or TAU, and nested patients within clinician intervention status.

Patients were recruited via mailings and advertising flyers; those with chart-documented musculoskeletal pain diagnoses who reported at least moderate pain severity and pain-related function (Chronic Pain Grade [CPG]) lasting at least 12 weeks were invited to participate. Participants completed questionnaires at baseline, 3, 6 and 12 months, with a subset re-assessed at 30 months. Primary outcomes were Roland-Morris Disability scores and CPG pain intensity scale scores over 12 months. Depression was assessed using Patient Health Questionnaire 9 [PHQ-9] scores. Intervention effects on patient outcome variables were tested using intention-to-treat analyses with multilevel models; patient-level covariates of age, sex, baseline depression severity, baseline opioid status (yes/no), and medical morbidity were included. To quantify provider adherence to pain treatment guidelines, we created the Pain Process Measure (PPM), a chart review checklist. Clinicians completed a baseline 23-item survey of attitudes and behaviors related to chronic pain management, job satisfaction, and satisfaction with local pain resources. Patient satisfaction measures included patient-rated global impression of change, global VA health care satisfaction, health-related quality of life, and receipt and rating of effectiveness of VA chronic pain treatment. Pain disability-free days were calculated from Roland-Morris Disability Questionnaire scores. Data on VA treatment costs were obtained from the VA's Decision Support System for all utilization except certain intervention activities that were tracked in a separate study database.

Status:

Complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently receiving primary care at Portland VAMC
* Diagnosed musculoskeletal chronic pain condition lasting at least 3 months
* Currently experiencing moderate to severe symptoms as per screening
* Willingness to complete 6 and 12 month interviews
* Regular access to a telephone

Exclusion Criteria:

* Dementia or cognitive disturbance
* Diagnoses of fibromyalgia, chronic fatigue or somatization disorder Terminal illness
* Designated guardian
* Drug-seeking behavior flag in medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Dobscha, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

REFERENCES:
- [Background] Otis JD, Macdonald A, Dobscha SK. Integration and coordination of pain management in primary care. J Clin Psychol. 2006 Nov;62(11):1333-43. doi: 10.1002/jclp.20313. PMID 16937344
- [Result] Dobscha SK, Corson K, Perrin NA, Hanson GC, Leibowitz RQ, Doak MN, Dickinson KC, Sullivan MD, Gerrity MS. Collaborative care for chronic pain in primary care: a cluster randomized trial. JAMA. 2009 Mar 25;301(12):1242-52. doi: 10.1001/jama.2009.377. PMID 19318652
- [Result] Morasco BJ, Dobscha SK. Prescription medication misuse and substance use disorder in VA primary care patients with chronic pain. Gen Hosp Psychiatry. 2008 Mar-Apr;30(2):93-9. doi: 10.1016/j.genhosppsych.2007.12.004. PMID 18291290
- [Result] Dobscha SK, Corson K, Leibowitz RQ, Sullivan MD, Gerrity MS. Rationale, design, and baseline findings from a randomized trial of collaborative care for chronic musculoskeletal pain in primary care. Pain Med. 2008 Nov;9(8):1050-64. doi: 10.1111/j.1526-4637.2008.00457.x. Epub 2008 Jun 18. PMID 18565008
- [Result] Dobscha SK, Leibowitz RQ, Flores JA, Doak M, Gerrity MS. Primary care provider preferences for working with a collaborative support team. Implement Sci. 2007 May 30;2:16. doi: 10.1186/1748-5908-2-16. PMID 17537251
- [Result] Dickinson KC, Sharma R, Duckart JP, Corson K, Gerrity MS, Dobscha SK. VA healthcare costs of a collaborative intervention for chronic pain in primary care. Med Care. 2010 Jan;48(1):38-44. doi: 10.1097/MLR.0b013e3181bd49e2. PMID 19952802
- [Result] Morasco BJ, Dobscha SK. Impact of comorbid substance use disorder on pain functioning: 12-month follow-up evaluation. [Abstract]. Annals of behavioral medicine : a publication of the Society of Behavioral Medicine. 2010 Apr 1; 39(Suppl):S185.
- [Result] Morasco BJ, Corson K, Turk DC, Dobscha SK. Association between substance use disorder status and pain-related function following 12 months of treatment in primary care patients with musculoskeletal pain. J Pain. 2011 Mar;12(3):352-9. doi: 10.1016/j.jpain.2010.07.010. Epub 2010 Sep 20. PMID 20851057
- [Result] Morasco BJ, Gritzner S, Lewis L, Oldham R, Turk DC, Dobscha SK. Systematic review of prevalence, correlates, and treatment outcomes for chronic non-cancer pain in patients with comorbid substance use disorder. Pain. 2011 Mar;152(3):488-497. doi: 10.1016/j.pain.2010.10.009. Epub 2010 Dec 23. PMID 21185119
- [Result] Dobscha SK, Corson K, Flores JA, Tansill EC, Gerrity MS. Veterans affairs primary care clinicians' attitudes toward chronic pain and correlates of opioid prescribing rates. Pain Med. 2008 Jul-Aug;9(5):564-71. doi: 10.1111/j.1526-4637.2007.00330.x. PMID 18777608
- [Result] Denneson LM, Corson K, Dobscha SK. Complementary and alternative medicine use among veterans with chronic noncancer pain. J Rehabil Res Dev. 2011;48(9):1119-28. doi: 10.1682/jrrd.2010.12.0243. PMID 22234716
- [Result] Morasco BJ, Duckart JP, Dobscha SK. Adherence to clinical guidelines for opioid therapy for chronic pain in patients with substance use disorder. J Gen Intern Med. 2011 Sep;26(9):965-71. doi: 10.1007/s11606-011-1734-5. Epub 2011 May 12. PMID 21562923
- [Result] Corson K, Doak MN, Denneson L, Crutchfield M, Soleck G, Dickinson KC, Gerrity MS, Dobscha SK. Primary care clinician adherence to guidelines for the management of chronic musculoskeletal pain: results from the study of the effectiveness of a collaborative approach to pain. Pain Med. 2011 Oct;12(10):1490-501. doi: 10.1111/j.1526-4637.2011.01231.x. Epub 2011 Sep 21. PMID 21943325
- [Result] Thielke S, Corson K, Dobscha SK. Collaborative care for pain results in both symptom improvement and sustained reduction of pain and depression. Gen Hosp Psychiatry. 2015 Mar-Apr;37(2):139-43. doi: 10.1016/j.genhosppsych.2014.11.007. Epub 2014 Nov 21. PMID 25554014

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: Pain treatment as usual
Period: Overall Study
Arm/Group | Assistance With Pain Treatment | Treatment as Usual
Started | 187 | 214
Completed | 187 | 214
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Veterans receiving healthcare in VA primary care
Groups:
- Treatment as Usual: Treatment as usual which includes standard pain care, clinician generated referrals for additional consultation and ancillary services
- Total: Total of all reporting groups
Arm/Group | Assistance With Pain Treatment | Treatment as Usual | Total
Number analyzed (Participants) | 187 | 214 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (12.3) | 62.1 (11.2) | 61.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 172 | 196 | 368
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 168 | 189 | 357
  Black | 2 | 5 | 7
  American Indian/Alaska Native | 7 | 6 | 13
  Unknown | 10 | 14 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 187 | 214 | 401

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Change in Pain-related Function (Roland Disability Score)
Description: The Roland Morris Disability Questionnaire has 24 yes or no items. Each item is scored as 0 or 1. Item scores or summed to create total score with range 0 to 24. Higher scores represent greater disability. The Roland Morris has been widely used, has content and construct validity, internal consistency, and responsiveness to change among patients with chronic pain.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Assistance With Pain Treatment (Intervention): Care management intervention including assessment, decision support, patient activation, education and followup, provider education, feedback to providers
  Assistance with Pain treatment: Care management intervention including assessment, decision support, patient activation, education and followup, provider education, feedback to providers. Intervention delivered for 12 months.
Arm/Group | Assistance With Pain Treatment (Intervention) | Treatment as Usual
Number analyzed (Participants) | 187 | 214
units on a scale | -1.4 [-2.0 to -.71] | -0.2 [-0.8 to 0.4]

2. Secondary Outcome: Adjusted Change in Depression Severity
Description: Patient Health Questionnaire-9 depression rating scale. Range 0-27 with higher scores representing higher depression severity
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Assistance With Pain Treatment (Intervention) | Treatment as Usual
Number analyzed (Participants) | 187 | 214
units on a scale | -3.7 [-4.9 to -0.24] | -1.2 [-4.9 to -0.24]

3. Secondary Outcome: Adjusted Change in Pain Interference
Description: Chronic Pain Grade interference score. Range 0 to 100 with higher scores representing greater pain interference (worse outcome)
Time Frame: 12 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Assistance With Pain Treatment (Intervention) | Treatment as Usual
Number analyzed (Participants) | 187 | 214
units on a scale | -5.7 [-9.8 to -1.7] | 2.3 [-1.6 to 6.1]

4. Secondary Outcome: Global Impression of Change
Description: Global impression of change score. Rated at 12 months capturing patient impression of change over past 6 months. Range 1-7 with lower scores representing greater improvement
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Assistance With Pain Treatment (Intervention) | Treatment as Usual
Number analyzed (Participants) | 187 | 214
units on a scale | 3.7 [3.5 to 3.8] | 4.4 [4.3 to 4.6]

5. Secondary Outcome: Adjusted Change in Health Related Quality of Life
Description: EQ-5D. Range 3-15 with higher scores representing worse health states
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Assistance With Pain Treatment (Intervention) | Treatment as Usual
Number analyzed (Participants) | 187 | 214
units on a scale | -0.02 [-0.05 to 0.01] | -0.04 [-0.05 to -0.02]

ADVERSE EVENTS:
Groups:
- Treatment as Usual: Treatment as usual, which includes standard pain care, clinician-generated referrals for additional consultation and ancillary services
Arm/Group | Assistance With Pain Treatment | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/187 | 0/214
Other Adverse Events (participants affected / at risk) | 0/187 | 0/214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes